CLINICAL TRIAL: NCT06675071
Title: Mortality Risk Assessment by Skilled Staff Compared to Existing Validated Tools in Skilled Nursing Departments
Status: Not yet recruiting | Type: Observational
Sponsor: Shmuel Harofeh Hospital, Geriatric Medical Center (Other Government)
Responsible Party: Principal Investigator, Yochai Levy, Hospital deputy director, Shmuel Harofeh Hospital, Geriatric Medical Center
Other Study IDs: SH-118-24
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Mortality Prediction
Keywords: older adults, long term care, Mortality Prediction; MITCHELL scale, POROCK scale

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Mortality Risk Assessment by Skilled Caregivers Compared to Existing Validated Tools in Skilled Nursing Departments at Shmuel Harofeh Geriatric Hospital

Background The elderly population in Israel and globally is growing, increasing demand for medical services, particularly palliative care. Recommendations from 2016 emphasized the need for geriatric and skilled nursing departments to focus on end-of-life care, but implementation has been limited. High mortality and frequent readmissions are reported in long-term care, yet accurate mortality prediction tools for elderly patients remain limited. Improved mortality prediction can help identify patients who would benefit from palliative care and reduce unnecessary interventions.

Research Objectives

1. Assess life expectancy of patients in skilled nursing departments.
2. Compare the effectiveness of various tools in predicting six-month mortality.

Hypothesis Caregiver assessments will more accurately predict mortality than current validated tools.

Study Design Type: Prospective cohort study. Location: Shmuel Harofeh Hospital

Study Population Approximately 250 patients admitted to skilled nursing departments at Shmuel Harofeh Hospital.

Recruitment Period: Two years. Follow-up Period: Up to one year.

Methods

Epidemiological and clinical data (age, comorbidities, functional and cognitive status, lab results) will be collected. Mortality risk will be assessed using:

1. Validated Tools: Including the MITCHELL scale (for patients with advanced dementia) and the POROCK scale (for institutionalized patients).
2. Caregiver Assessment: Subjective life expectancy estimates by attending geriatricians and nursing staff within three days of admission and again 7-10 days later. An external geriatrician will also provide an assessment based on brief, non-invasive observation.

Data Processing Data will be coded, entered into an electronic dataset, and undergo statistical analysis after collection. No interventions beyond routine care are included.

Ethical Considerations As an observational study without intervention, a waiver for informed consent was granted.

Importance of Research Skilled nursing facilities increasingly need to provide palliative care for elderly patients. This study aims to improve mortality prediction methods, helping to identify patients for end-of-life care, ultimately enhancing care quality, and reducing costs by avoiding unnecessary hospitalizations and treatments.

ELIGIBILITY:
Inclusion Criteria: Patients admitted to skilled nursing departments at Shmuel Harofeh Hospital.

-

Exclusion Criteria: Patients admitted for end-of-life care

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients over the age of 65 years admitted to skilled nursing departments at Shmuel Harofeh Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-11-10 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
life expectancy of patients in skilled nursing departments | 3 years
  Compare the effectiveness of various tools in predicting six-month mortality

IPD SHARING:
Plan to Share IPD: No